CLINICAL TRIAL: NCT05714124
Title: Liver Embolization Approaches for Tumor Management - Retrospective and Prospective Analysis of the Short-, Medium-, and Long-term Clinical Course of Patients Subjected to Embolization Treatment for Primary and Secondary Liver Neoplasms
Brief Title: Liver Embolization Approaches for Tumor Management
Acronym: LEATUM
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco De Cobelli, Head of Radiology, IRCCS San Raffaele
Other Study IDs: LEATUM
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma; Metastatic Colon Cancer; Metastatic Cancer; Metastatic Gastric Cancer; Primary Liver Cancer; Metastatic Pancreatic Cancer
Keywords: embolization, TAE, TACE, TARE, PVE, HVE
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Colonic Neoplasms; Neoplasm Metastasis; Stomach Neoplasms; Pancreatic Neoplasms | interventions — Embolization, Therapeutic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Embolization — Endovascular treatment for patients with primary and secondary liver tumors
  Other Names: Transarterial Chemoembolisation; Transarterial Radioembolization; Bland Transarterial Embolization; Hepatic Vein Embollization; Portal Vein Embolization

SUMMARY:
The goal of this evaluate short, medium and long term outcome of the different embolization techniques in patients with primary and secondary hepatic tumors. The main aim is to evaluate progression free survival following embolization in this study population or evaluate residual hepatic volume in cases in which these techniques are used to induce liver regeneration. This study is an observational registry - all patients will follow their normal therapeutic and treatment scheme as per clinical practice, without any additional intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 yoa
* patients with patients with primary or secondary liver disease not amenable for surgery or ablation
* patients with primary or secondary liver tumors candidates for major surgery prior to induction of hypertrophy
* able and willing to sign informed consent

Exclusion Criteria:

* pregnant women
* patients with uncorrectable coagulopathy
* diffuse extrahepatic disease
* for lobar TACE and TARE - presence of bilodigestive shunt
* for TARE - >20% hepatopulmonary shunt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or secondary liver tumors
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Short term (3-6 months)
  Treatment Efficacy
Progression free survival | From time of intervention up to 1 year (medium term)
Progression free survival | From time of intervention up to 5 years (Long term)
Residual hepatic volume | within 40 days of procedure
  Treatment Efficacy

SECONDARY OUTCOMES:
Overall survival | From date of procedure until the date of death from any cause, whichever came first, assessed up to 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy